CLINICAL TRIAL: NCT06483282
Title: A Single-arm, Prospective, Exploratory Study of Adebrelimab Combined With Apatinib Mesylate and Chemotherapy for Neoadjuvant Therapy and Biomarker Analysis in Limited-stage Small Cell Lung Cancer
Brief Title: A Study of Adebrelimab Combined With Apatinib Mesylate and Chemotherapy for Neoadjuvant Therapy and Biomarker Analysis in Limited-stage Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jin Ying (Other)
Responsible Party: Sponsor-Investigator, Jin Ying, Associate chiefphysician, Department of Thoracic Medicine, Zhejiang Cancer Hospital
Organization: Zhejiang Cancer Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2024-420
Record Dates: First submitted 2024-05-23; First posted 2024-07-03 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Small Cell Lung Cancer Limited Stage
MeSH Terms: interventions — apatinib; Etoposide; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adebrelimab in combination with chemotherapy and apatinib mesylate (Experimental): Adebrelimab 1200mg q3w for 4 cycles, Apatinib mesylate 250mg qod q3w 3 times/week concurrent with adebrelimab for 3 cycles, platinum-based chemotherapy (etoposide, 100mg/m2, q3w; Carboplatin, AUC=5, q3w), 4 cycles, and operation was performed within 4-8 weeks after treatment (Apatinib mesylate was discontinued for 4 weeks). According to the results of MDT discussion, adebrelimab, 1200mg q3w, and apatinib 250mg qod q3w 3 times/week were used 4 weeks after surgery, which with or without radiotherapy. Preoperative prophylactic radiotherapy (PCI) is recommended for patients with preoperative stage N1. Patients with postoperative stage N1 received postoperative thoracic radiotherapy.
  Interventions: Drug: Adebrelimab; Drug: Apatinib Mesylate; Drug: Etoposide; Drug: Carboplatin

INTERVENTIONS:
Drug: Adebrelimab — This product is administered by intravenously guttae. The recommended dose of subcutaneous injection is 20mg/kg, administered every 3 Weeks (Q3W).
  Other Names: SHR-1316
Drug: Apatinib Mesylate — This product is an orally administered targeted therapy drug, with a recommended dosage of one tablet per day.
Drug: Etoposide — This product is administered by intravenously guttae. The recommended dose of subcutaneous injection is 100mg/m2, administered every 3 Weeks (Q3W).
Drug: Carboplatin — This product is administered by intravenously guttae. AUC=5, administered every 3 Weeks (Q3W).

SUMMARY:
This is a single-arm, prospective, exploratory phase II clinical study. The study enrolled newly diagnosed stage T1-3N0-1M0 resectable limited-stage small cell lung cancer. Adebrelimab combined with chemotherapy for 4 cycles and apatinib mesylate for 3 cycles. Surgery was performed within 4-8 weeks after the above treatment (the operation was performed 4 weeks after apatinib was discontinued). According to the results of MDT discussion, adebrelimab combined with apatinib mesylate combined with or without radiotherapy was started 4 weeks after surgery. Preoperative prophylactic radiotherapy (PCI) is recommended for patients with preoperative stage N1. Patients with postoperative stage N1 received postoperative thoracic radiotherapy.

DETAILED DESCRIPTION:
Preoperative prophylactic radiotherapy (PCI) is recommended for patients with preoperative stage N1. Patients with postoperative stage N1 received postoperative thoracic radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years old;
* Histologically or cytologically confirmed limited-stage small cell lung cancer (T1-3N0-1M0).
* All lesions of the patient (including the primary lesion, lymph nodes/lesions assessed as metastatic) must be jointly evaluated and confirmed as resectable by a surgeon, a radiation oncologist, and a radiologist;
* The subject must have measurable target lesions (according to RECIST 1.1 criteria);
* ECOG performance status score of 0-1;
* No history of other malignancies;
* No previous treatment for small cell lung cancer-related surgery, radiotherapy, chemotherapy, immunotherapy, or other anti-tumor treatments;
* The patient must have adequate cardiopulmonary function: the patient's FEV1 and DLCO are both ≥50% of the predicted value, echocardiography shows LVEF ≥55%, and no clear signs of heart failure, severe coronary artery stenosis, etc., are seen on various tests, and the cardiopulmonary function is assessed by a surgeon as being able to tolerate surgical treatment;
* The levels of important organ functions must meet the following requirements: a. Bone marrow: Absolute neutrophil count (ANC) ≥1.5×10^9/L, platelets ≥100×10^9/L, hemoglobin ≥9 g/dl; b. Good coagulation function: defined as international normalized ratio (INR) or prothrombin time (PT) ≤1.5 times the upper limit of normal (ULN); c. Liver: Total bilirubin ≤1.5 times the upper limit of normal, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 times the upper limit of normal; d. Kidney: Serum creatinine ≤1.25 times the upper limit of normal or creatinine clearance (calculated using the Cockcroft-Gault formula) ≥60 ml/min;
* Males with reproductive capacity and women of childbearing age must agree to use effective contraception from the time of signing the main informed consent form until 180 days after the last administration of the study drug. Women of childbearing age include pre-menopausal women and post-menopausal women within 2 years. The pregnancy test result of women of childbearing age must be negative within ≤7 days before the first administration of the study drug;
* Voluntarily participate in clinical research; fully understand and be informed about this study and sign the informed consent form.

Exclusion Criteria:

* Inability to completely remove all lesions through surgery;
* Received anti-tumor treatment for SCLC (including but not limited to chemotherapy, radiotherapy of the lesion area).
* Previously used immunocheckpoint inhibitors such as PD-1/PD-L1 inhibitors for treatment.
* Any history of active autoimmune diseases or autoimmune diseases (such as uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism (can be included after hormone replacement therapy), tuberculosis); patients with childhood asthma that has completely resolved and does not require any intervention in adulthood or vitiligo can be included, but patients requiring medical intervention with bronchodilators are not eligible for inclusion;
* Have congenital or acquired immune system deficiencies, such as human immunodeficiency virus (HIV) infected individuals, active hepatitis B (HBV DNA ≥ 500 IU/ml), hepatitis C (positive for hepatitis C antibodies and HCV-RNA is above the lower limit of detection of the analytical method) or co-infection with both hepatitis B and C;
* Existence of uncontrollable third-space effusions, such as a large amount of pleural effusion or ascites or pericardial effusion;
* Subjects who need systemic treatment with corticosteroids (>10 mg/day prednisone or equivalent) or other immunosuppressants within 14 days before the first administration of the drug. Inhaled or topical corticosteroids are allowed, as well as adrenal hormone replacement therapy with a dose >10 mg/day prednisone equivalent, in the absence of active autoimmune diseases;
* Subjects who have been treated with anti-tumor vaccines or other immunostimulatory anti-tumor drugs (interferons, interleukins, thymosin, immune cell therapy, etc.) within 1 month before the first administration of the drug;
* Currently participating in other interventional clinical studies;
* Evidence of previous or current pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-induced pneumonia, and severe lung function impairment;
* Patients with severe heart disease, such as congestive heart failure grade III or above (NYHA standard), or angina grade III or above (CCS standard), or a history of myocardial infarction within 6 months before treatment initiation, or arrhythmias requiring drug treatment;
* Major surgery, open biopsy, or significant trauma within 28 days before enrollment;
* Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
* Pregnant or breastfeeding women; patients with fertility who are unwilling or unable to take effective contraceptive measures;
* Known allergic reactions, hypersensitivity, or intolerance to the study drug;
* Hypertension that cannot be well controlled with antihypertensive drug treatment (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg);
* Abnormal coagulation function (INR > 2.0 or prothrombin time (PT) > 16s), with a tendency to bleed or currently undergoing thrombolysis or anticoagulant treatment (preventive use of low-dose aspirin, low molecular weight heparin is allowed);
* Significant clinical bleeding symptoms within the last 3 months or a clear tendency to bleed, such as gastrointestinal bleeding, bleeding gastric ulcers, or patients with vasculitis, etc., if the baseline fecal occult blood is positive, it can be retested, and if it is still positive after retesting, an endoscopy is required (except for those who have undergone endoscopy within 3 months and before the baseline period to rule out such conditions);
* Arterial/venous thrombotic events within the last 6 months, such as cerebrovascular accidents (including transient ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism;
* Known genetic or acquired bleeding and thrombotic tendencies (such as hemophilia, coagulation disorders, thrombocytopenia, etc.). Other conditions deemed unsuitable for participating in the study by the researcher.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-06-21 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
EFS of 2 years | Up to 2 years
  The proportion of patients who did not experience any of the following events from the start of treatment to 2 years: disease progression without surgical treatment, local or distant recurrence, death from any cause, etc.

SECONDARY OUTCOMES:
MPR | Up to 2 years
  MPR (Major Pathological response,) was defined as residual tumor cells ≤10% in pathological examination of postoperative specimens.
EFS | Up to 2 years
  EFS (Event-Free Survival) refers to the time from the beginning of randomization to the first occurrence of any of the following events: disease progression without surgical treatment, local or distant recurrence, death from any cause, etc.
OS | Up to 2 years
  OS (Overall Survival), the time from the date of randomization until the death of the participant or the last follow-up.
ORR | Up to 2 years
  ORR (Objective Response Rate) refers to the proportion of patients whose tumor shrinkage reaches a certain level and remains for a certain period of time, including complete response (CR) and partial response (PR) cases.
Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to 2 years
  Number of participants with treatment-related adverse events as assessed by NCI-CTCAE v5.0.
pCR | Up to 2 years
  pCR, Pathological Complete Response, defined as the complete absence of all tumor cells in the primary site and lymph nodes.

CONTACTS AND LOCATIONS:
Overall Officials: Da Chen, MD&PhD, Study Chair — Medical Ethics Committee Of Zhejiang Cancer Hospital; Zhengfu He, MD&PhD, Principal Investigator — Sir Run Run Shaw Hospital; Zhengliang Tu, MD&PhD, Principal Investigator — Zhejiang University; Junqiang Fan, MD&PhD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No